CLINICAL TRIAL: NCT02330367
Title: Safety, Tolerability, Pharmacokinetics and Anti-tumour Activity of AC0010 in Patients With EGFR T790M Positive Advanced Non Small Cell Lung Cancer Who Progressed on Prior Therapy With EGFR TKIs
Brief Title: Safety, Pharmacokinetic and Preliminary Efficacy Study of AC0010 in Patients With EGFR T790M Positive NSCLC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hangzhou ACEA Pharmaceutical Research Co., Ltd. (Industry)
Collaborators: Guangdong Provincial People's Hospital (Other); Acea Bio (Hangzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC201410AVTN02.
Record Dates: First submitted 2014-12-31; First posted 2015-01-01 (Estimated); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Metastatic Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — abivertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AC0010 (Experimental): Oral AC0010 monotherapy
  Interventions: Drug: AC0010

INTERVENTIONS:
Drug: AC0010 — Phase 1: AC0010 will be administered in escalating dosages in a period of 28-day cycles.
  Phase 2: AC0010 will be administered twice-daily at RP2D.
  Other Names: AC0010MA

SUMMARY:
AC0010 is a novel, potent, small molecule irreversible tyrosine kinase inhibitor (TKI) that selectively targets mutant forms of the epidermal growth factor receptor (EGFR) while sparing wild-type (WT) EGFR. The purpose of the study is to evaluate the pharmacokinetic (PK) and safety profile of oral AC0010; to determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of oral AC0010; to assess the safety and efficacy of AC0010 in previously treated mutant EGFR in NSCLC patients with EGFR T790M mutation.

DETAILED DESCRIPTION:
Lung cancer remains the most common cancer worldwide with non-small cell lung cancer (NSCLC) accounting for 85% of cases. Molecularly targeted therapies have proven to be superior to chemotherapy for NSCLC patients whose tumors have mutations in EGFR. Recent studies have established tyrosine kinase inhibitors (TKIs) as the gold standard for treating EGFR-mutation-positive NCSLC. However, patients on TKIs eventually progress, and in approximately 50% of cases, progression is due to development of an additional mutation called T790M. AC0010 may provide an effective therapy for a patient population with few alternative treatment options. Pre-clinical data demonstrated that AC0010 inhibits T790M. It is anticipated that AC0010 may promote cell death in tumor cells with the T790M mutation, thus providing possible therapeutic benefit in patients who have developed T790M-mediated resistance to previous TKIs.

This is a two-part, open-label study of oral AC0010 administered twice-daily in previously treated NSCLC patients who have documented evidence of an activating mutation in the EGFR gene and have failed treatment with an EGFR inhibitor such as erlotinib, gefitinib or afatinib.

This study will include 2 parts:

phase 1 : Dose-escalation Period with 28-day cycles; Optional Treatment Extension Period starting on Day 29

phase 2 : Evaluation of activity and safety in patients with the EGFR T790M mutation

ELIGIBILITY:
Inclusion Criteria - phase 1:

1. Patients of either gender, aged from 18 years older to 75.
2. Histologically or cytologically confirmed metastatic, or unresectable locally advanced, recurrent NSCLC.
3. At least one measurable disease by CT or MRI, according to RECIST Version 1.1.
4. Failed to the treatment of EGFRTKI with definite state of T790M, or harbored T790M mutation without the treatment of EGFRTKI.
5. Offer biopsy sample to central lab if failed or without the treatment of EGFRTKI.
6. Adequate hematological and physiological functions of heart, lung, liver, and kidney according to definitions given in Appendix D.
7. Any prior treatment (including chemotherapy, radiotherapy, biotherapy and other clinical medicine) must be completed over 28 days or 5 half-lives from the screening.
8. ECOG (Eastern Cooperative Oncology Group) performance status of 0 to 1.
9. NSCLC patients with asymptomatic brain metastasis or drug-controllable brain metastasis.
10. Life expectancy of at least 3 months.
11. Patients should cooperate with investigator to observe adverse events and efficacy.
12. Without other anticancer therapy.
13. Women without pregnancy or breastfeeding.
14. Adequate function of blood coagulation (INR≤1.5)
15. Signed consent on an Independent Ethics Committee-approved Informed Consent Form prior to any study-specific evaluation.

Exclusion Criteria - Phase 1:

1. No pathology confirmation.
2. HCV positive, active hepatitis B.
3. History of interstitial lung disease related to prior EGFR inhibitor therapy.
4. Positive to HIV antibody or other immunodeficiency disease or organ transplantation.
5. Residue toxicity related to prior therapies > grade 1.
6. BUN or Cr > 1.5 × upper limits of normal.
7. ALT or AST > 2.5 × upper limits of normal, total bilirubin> 1.5 × upper limits of normal.
8. Fever (temperature>38℃ or any uncontrolled active infections.
9. Patients received high-dose glucocorticoid or any other immunosuppression within 1 month.
10. Any severe or uncontrolled disease, such as mental, neurologic, cardiovascular, respiratory diseases.
11. Patients with symptomatic and untreated brain metastasis.
12. Patients with organic heart disease, cardiac insufficiency, >2 degree heart block, experienced myocardial infarction in 6 months. Abnormal PR, QT, QRS interval (defined as: 12 lead electrocardiogram QT interval correlated to Bazetts (QTcB)>450ms (male) or >470ms (female), PR>240ms, QRS>110ms).
13. Patients receiving medication known to prolong QT interval.
14. Past history of major surgery in 14 days prior to enrollment.
15. Pregnant or lactating women.
16. Any other reasons for the investigator to consider the patient should not participate in the study.

Inclusion Criteria - Phase 2:

1. Patients of either gender, aged from 18 years older to 75.
2. Histologically or cytologically confirmed metastatic, or unresectable locally advanced, recurrent NSCLC.
3. At least one measurable disease by CT or MRI, according to RECIST Version 1.1.
4. Failed to the treatment of EGFR-TKI and harbored T790M mutation.
5. Offer biopsy sample to central lab if failed or without the treatment of EGFRTKI.
6. Patients failed the treatment of EGFR-TKI should be treated with only one kind of medicine. Patients with arbored T790M mutation should be treated with only one kind of medicine or never be treated.
7. Comply with the results of laboratory testing.
8. ECOG (Eastern Cooperative Oncology Group) performance status of 0 to 1 and no deterioration in 2 weeks.
9. Life expectancy of more than 12 weeks.
10. Patients should cooperate with investigator to observe adverse events and efficacy.
11. Women without pregnancy.
12. Signed consent on an Independent Ethics Committee-approved Informed Consent Form prior to any study-specific evaluation.

Exclusion Criteria - Phase 2:

1. Acute and chronic hepatitis C, active hepatitis B (including positive HBsAg and/or HBeAg; HBcAb and/or positive HBeAb and positive HBV DNA), hepatitis E Virus IgM antibody positive.
2. History of interstitial lung disease related to prior EGFR inhibitor therapy.
3. Positive to HIV antibody or other immunodeficiency disease or organ transplantation.
4. Fever (temperature>38℃ or any uncontrolled active infections.
5. Patients received high-dose glucocorticoid or any other immunosuppression within 1 month.
6. Any severe or uncontrolled disease, such as mental, neurologic, cardiovascular, respiratory diseases.
7. ECG showed abnormal rhythm, conduction and form, such as complete left bundle branch block, >2 degree heart block, PR interval >250ms, experienced myocardial infarction in 6 months. Risks leading to prolonged QT interval or arrhythmia, such as heart failure, hypokalemia, congenital long QT, long QT family history or sudden death under 40 years old in first degree relatives (12 lead electrocardiogram QT interval correlated to Bazetts (QTcB) > 450ms.
8. Prior history of malignancies other than NSCLC (except cured malignancy such as removed basal-cell carcinoma and carcinoma in situ) within 5 years.
9. Patients with CNS metastasis (except asymptomatic CNS metastasis with stable radiography in 4 weeks and no long-term use of corticosteroid. CNS metastasis focuses ≤2, maximum diameter of focus <10mm)
10. Radiation field covered more than 30% bone marrow within 4 weeks of enrollment.
11. Lab test of 1ml plasma prove treatment of AZD9291.
12. Patients already received treatment of this research or quite the treatment of this research. Patients treated with 3rd generation of EGFR-TKI (AZD9291, AC0010, BPI-15086, CO-1686, HM61713).
13. Past history of major surgery in 14 days prior to enrollment.
14. Pregnant or lactating women.
15. Patients with uncontrolled pleural effusion and/or pericardial effusion.
16. Any other reasons for the investigator to consider the patient should not participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
ORR(Objective Response Rate) | Every 6 weeks from time of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 11 months
  To assess the overall objective response rate (ORR) of AC0010 in EGFR T790M mutation-positive patients with advanced non-small cell lung cancer (NSCLC).

SECONDARY OUTCOMES:
DoR (Duration of Response) | Every 6 weeks from time of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 11 months
  To assess the duration of response (DOR) of AC0010 in EGFR T790M mutation-positive patients with advanced non-small cell lung cancer (NSCLC).
PFS (Progression-free survival) | Every 6 weeks from time of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 11 months
  To assess the progression-free survival (PFS) of AC0010 in EGFR T790M mutation-positive patients with advanced non-small cell lung cancer (NSCLC).
DCR (Disease control rate) | Every 6 weeks from time of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 11 months
  To assess the disease control rate (DCR) of AC0010 in EGFR T790M mutation-positive patients with advanced non-small cell lung cancer (NSCLC).
OS (Overall survival) | Every 6 weeks from time of first dose until objective disease progression, then every 3 months until death of lost of follow-up, up to approximately 18 months
  To assess the overall survival (OS) of AC0010 in EGFR T790M mutation-positive patients with advanced non-small cell lung cancer (NSCLC).
EORTC QLQ-C30 and LC-13 questionnaire | From screening to the end of survival follow-up, which is assessed though study completion
  To assess the safety of AC0010 in EGFR T790M mutation-positive patients with advanced non-small cell lung cancer (NSCLC).
Adverse events | From screening to 30days after end of treatment, which is assessed through study completion
  To assess the safety of AC0010 in EGFR T790M mutation-positive patients with advanced non-small cell lung cancer (NSCLC).

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wu, MD., Principal Investigator — Guangdong Provincial People's Hospital
Locations (17):
- China (17):
  - 307 Hospital of PLA, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nanjing General Hospital of Nanjing Military Command, Nanjing, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - West China Hospital,Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hanzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang YC, Chen ZH, Zhang XC, Xu CR, Yan HH, Xie Z, Chuai SK, Ye JY, Han-Zhang H, Zhang Z, Bai XY, Su J, Gan B, Yang JJ, Li WF, Tang W, Luo FR, Xu X, Wu YL, Zhou Q. Analysis of resistance mechanisms to abivertinib, a third-generation EGFR tyrosine kinase inhibitor, in patients with EGFR T790M-positive non-small cell lung cancer from a phase I trial. EBioMedicine. 2019 May;43:180-187. doi: 10.1016/j.ebiom.2019.04.030. Epub 2019 Apr 23. PMID 31027916
- [Derived] Wang H, Zhang L, Hu P, Zheng X, Si X, Zhang X, Wang M. Penetration of the blood-brain barrier by avitinib and its control of intra/extra-cranial disease in non-small cell lung cancer harboring the T790M mutation. Lung Cancer. 2018 Aug;122:1-6. doi: 10.1016/j.lungcan.2018.05.010. Epub 2018 May 21. PMID 30032814